CLINICAL TRIAL: NCT05818033
Title: Safety and Effectiveness of CARE1.02 Spectacle Lens Versus Single-vision Spectacle Lens in Myopia Control: a Randomised Controlled Trial
Brief Title: Safety and Effectiveness of CARE1.02 Spectacle Lens in Myopia Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023KYPJ005
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-03

CONDITIONS: Myopia
Keywords: Myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): CARE1.02
  Interventions: Device: CARE1.02
- Control group (Active Comparator): Single-vision spectacle lens
  Interventions: Device: Single-vision spectacle lens

INTERVENTIONS:
Device: CARE1.02 — Participants in the intervention group will wear CARE1.02 and receive the follow-up checks.
  Arms: Intervention group
Device: Single-vision spectacle lens — Participants in the control group will wear single-vision spectacle lens and receive the follow-up checks.
  Arms: Control group

SUMMARY:
China is a major country in myopia, with the highest number of teenagers suffering from myopia. Controlling the progression of myopia and the related complications caused by axial elongation have clinical significance and social value. Currently. There is a lack of researches on the impact of specially designed myopia control spectacle lens in adolescents aged 12 and above. Therefore, The researchers plan to conduct a randomized controlled trial among myopia adolescents aged 12-17 in middle and high schools in Guangzhou, to test and verify the safety and effectiveness of CARE1.02 on myopia control compared with single-vision spectacle lens.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 17 years;
* Under the condition of bilateral cycloplegic autorefraction, the spherical refractive error of -0.50 to -8.00 D in each eye and astigmatism of not more than 1.50 D and anisometropia of not more than 1.50 D;
* Best-corrected visual acuity of equal or better than 0.00 LogMAR (>= 1.0 as Snellen).
* The intraocular pressure of 10 to 21mmHg.
* Volunteer to participate in this clinical trial with signature of the informed consent form.

Exclusion Criteria:

* History of eye injury or intraocular surgery;
* Clinically abnormal slit-lamp findings;
* Abnormal fundus examination;
* Ocular disease, such as uveitis and other inflammatory diseases,glaucoma, cataract, fundus diseases, eye tumors, dominant strabismus, and any eye diseases that affect visual function;
* Systemic diseases causing low immunity (such as diabetes, Down's syndrome, rheumatoid arthritis, psychotic patients or other diseases that researchers think are not suitable for wearing glasses);
* Participation of the drug clinical trial within three month and the device clinical trial within one month;
* Only one eye meets the inclusion criteria;
* Unable to have regular follow-up;
* Participation of any myopia control clinical research trial within three months, and currently using rigid contact lenses (including nursing products), multifocal contact lenses, progressive multifocal lenses and other specially designed myopia control lenses, atropine drugs, etc.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 760 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of spherical equivalent refraction (SER) at one year | 1 year
  The difference of SER at one year from baseline. SER will be measured after cycloplegia

SECONDARY OUTCOMES:
Changes of axial length (AL) at one year | 1 year
  The difference of AL at one year from baseline.
Change of anterior chamber depth (ACD) at one year | 1 year
  The difference of ACD at one year from baseline.
Change of lens thickness (LT) at one year | 1 year
  The difference of LT at one year from baseline.
Change of corneal curvature (CR) at one year | 1 year
  The difference of CR at one year from baseline.
Best corrected visual acuity at one year | 1 year
  Best corrected visual acuity
Binocular visual function at one year | 1 year
  Binocular visual function
Choroidal thickness at one year | 1 year
  The difference of Choroidal thickness at one year from baseline.
Visual scale score at 1 year | 1 year
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2)
Time length of wearing spectcales at one year | 1 year
  Time length of wearing spectcales collected every half year
Safty of wearing the spectacle lens | 1 year
  Safty of wearing the spectacle lens which is a qualitative outcome will be evaluated every half year by prespecified measures and definations through symptoms and signs, intraocular pressure#slit lamp and ocular fundus checks.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchs will share the IPD as request in future.

REFERENCES:
- [Background] Irving EL, Yakobchuk-Stanger C. Myopia progression control lens reverses induced myopia in chicks. Ophthalmic Physiol Opt. 2017 Sep;37(5):576-584. doi: 10.1111/opo.12400. Epub 2017 Jul 26. PMID 28746982
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Result] Naidoo KS, Fricke TR, Frick KD, Jong M, Naduvilath TJ, Resnikoff S, Sankaridurg P. Potential Lost Productivity Resulting from the Global Burden of Myopia: Systematic Review, Meta-analysis, and Modeling. Ophthalmology. 2019 Mar;126(3):338-346. doi: 10.1016/j.ophtha.2018.10.029. Epub 2018 Oct 17. PMID 30342076
- [Result] Wildsoet CF, Chia A, Cho P, Guggenheim JA, Polling JR, Read S, Sankaridurg P, Saw SM, Trier K, Walline JJ, Wu PC, Wolffsohn JS. IMI - Interventions Myopia Institute: Interventions for Controlling Myopia Onset and Progression Report. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M106-M131. doi: 10.1167/iovs.18-25958. PMID 30817829
- [Result] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039
- [Result] Smith EL 3rd, Hung LF. The role of optical defocus in regulating refractive development in infant monkeys. Vision Res. 1999 Apr;39(8):1415-35. doi: 10.1016/s0042-6989(98)00229-6. PMID 10343811
- [Result] Wallman J, Gottlieb MD, Rajaram V, Fugate-Wentzek LA. Local retinal regions control local eye growth and myopia. Science. 1987 Jul 3;237(4810):73-7. doi: 10.1126/science.3603011.
- [Result] Tse DY, Lam CS, Guggenheim JA, Lam C, Li KK, Liu Q, To CH. Simultaneous defocus integration during refractive development. Invest Ophthalmol Vis Sci. 2007 Dec;48(12):5352-9. doi: 10.1167/iovs.07-0383. PMID 18055781
- [Result] Arumugam B, Hung LF, To CH, Sankaridurg P, Smith EL III. The Effects of the Relative Strength of Simultaneous Competing Defocus Signals on Emmetropization in Infant Rhesus Monkeys. Invest Ophthalmol Vis Sci. 2016 Aug 1;57(10):3949-60. doi: 10.1167/iovs.16-19704. PMID 27479812
- [Result] Tse DY, To CH. Graded competing regional myopic and hyperopic defocus produce summated emmetropization set points in chick. Invest Ophthalmol Vis Sci. 2011 Oct 17;52(11):8056-62. doi: 10.1167/iovs.10-5207. PMID 21911586
- [Result] Woods J, Guthrie SE, Keir N, Dillehay S, Tyson M, Griffin R, Choh V, Fonn D, Jones L, Irving E. Inhibition of defocus-induced myopia in chickens. Invest Ophthalmol Vis Sci. 2013 Apr 12;54(4):2662-8. doi: 10.1167/iovs.12-10742. PMID 23471891